CLINICAL TRIAL: NCT01549158
Title: Randomized, Open-Label, Blinded-Endpoint, Crossover, Single Dose Study to Compare the Pharmacodynamics of Torasemide-PR 10 mg,Torasemide-IR 10 mg and Furosemide-IR 40 mg, in Patients With Compensated Heart Failure (CHF).
Brief Title: Single Dose Study to Compare the Pharmacodynamics of Torasemide-PR 10 mg,Torasemide-IR 10 mg and Furosemide-IR 40 mg in Patients With Compensated Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-110875-01
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Compensated Heart Failure
Keywords: loop diuretics; torasemide prolonged release; torasemide immediate release; Sutril Neo; pharmacodynamic profile of Torasemide-PR

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Torasemide PR 10 mg (Experimental)
  Interventions: Drug: torasemide-PR
- Furosemide-IR 40 mg (Active Comparator)
  Interventions: Drug: Furosemide-IR
- Torasemide-IR 10 mg (Active Comparator)
  Interventions: Drug: torasemide-IR

INTERVENTIONS:
Drug: torasemide-PR — Single oral dose of torasemide PR 10 mg
  Arms: Torasemide PR 10 mg
Drug: Furosemide-IR — Single oral dose of furosemide IR 40 mg
  Arms: Furosemide-IR 40 mg
Drug: torasemide-IR — Single oral dose of torasemide IR 10 mg
  Arms: Torasemide-IR 10 mg

SUMMARY:
This is a randomized, open-label, blinded-endpoint, crossover, single dose study to compare the pharmacodynamics of Torasemide-PR 10 mg, Torasemide-IR10 mg and furosemide-IR 40 mg. 30 patients of both sexes with CHF with a maximum imbalance of 60:40% in either direction will be included in the study. Patients with compensated heart failure, grade II or III as defined by the European Society of Cardiology, with a duration of ≥ 3 months at the time of inclusion documented in the patient's record or patients who previously required diuretic therapy.

Principal variable will be the efficiency of sodium excretion that will be assessed as the ratio between the average drug-induced natriuresis and the average drug recovered in urine over 24 hours.

The difference between the efficiency of 24 hour sodium excretion following administration of torasemide PR and furosemide will be formally tested by means of a Students t-test for paired samples. The test will be two-sided at 5% significance level. Efficiency changes over time will also be assessed, however will not be subject to formal statistical testing.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the nature of the study.
2. Obtain signed informed consent form approved by the Ethics Committee of the hospital (CEIC).
3. Male and female, ≥ 18 years at the time of the informed consent signature.
4. Patients with compensated heart failure, grade II or III as defined by the European Society of Cardiology, with a duration of ≥ 3 months at the time of inclusion documented in the patient's record or patients who previously required diuretic therapy.
5. Patients with stable heart failure on drug therapy. Stable drug therapy is defined as not having introduced any new drug for heart failure within 4 weeks prior to inclusion. Drugs doses could be adjusted during the study with the exception of the diuretics
6. Lab analysis results, vital signs and ECG within normal ranges or not considered clinically significant by the investigator.
7. For women only, the patient must be:

   * postmenopausal (≥ 1 year) or sterilized or,
   * without risk of becoming pregnant, not lactating, have a negative pregnancy test at study entry and without intention of becoming pregnant during the study course and use effective contraception.

   Postmenopausal status is defined as 12 consecutive months of spontaneous amenorrhea or confirmed by the results of follicle stimulating hormone (FSH) > 40 mlU/mL or at least 6 months after oophorectomy (with or without hysterectomy) documented in the patients record.
8. Body weight within the normal ranges (Quetelet's index between 19 and 30) expressed as weight (kg) /height (m2).

Exclusion Criteria:

1. Hospitalization due to heart failure, acute coronary syndrome, myocardial infarction, cardiac catheterization, revascularization, cardiac arrhythmia, transient ischemic attack or stroke, cardiac arrhythmia within 6 weeks prior to inclusion or major surgery including cardiac thoracic or within 8 weeks prior to inclusion.
2. Symptoms of angina at rest or with minimal activity (class III or IV, Canadian Cardiovascular Society).
3. Severe aortic or mitral stenosis or clinically significant valvular heart disease that can lead to surgery within 12 months after inclusion.
4. Hypertrophic obstructive cardiomyopathy, active myocarditis, constrictive pericarditis or clinically significant congenital heart disease.
5. If ventricular assist devices, continuous inotropic therapy or hospitalization is considered necessary in case of refractory end-stage heart failure.
6. Implementation of CRT within 3 months or cardioverter defibrillator in the 4 weeks before inclusion.
7. High probability of receiving a heart transplant within 6 months after inclusion.
8. Main organ transplant (ex. lungs, liver, kidney, heart, bone).
9. Positive surface antigen of hepatitis B, hepatitis C or HIV or a known diagnosis of AIDS.
10. Medical history or evidence of drug or alcohol abuse in the 3 months prior to inclusion.
11. Concomitant cardiovascular disease that is expected to reduce life expectancy to less than one year.
12. Scheduled routine iv infusions for heart failure (ex. inotropes, vasodilators, diuretics) or routine ultrafiltration.
13. Digoxin therapy at steady state (approximately 6 hours post-dose) exceeding 1.0 ng/mL at inclusion.
14. Chronic therapy with antiarrhythmic, antiepileptic drugs, eplerenone and espironolactone except amiodarone and beta-blockers.
15. Current intake or within 14 days prior to inclusion of a potent inhibitor of CYP2C9
16. Current intake or within 28 days prior to inclusion of a potent inducer of CYP2C9.
17. Participation, in the 60 days or 5 half lives preceding the inclusion in the study, in other clinical trial.
18. Systolic blood pressure > 150mm Hg diastolic blood pressure > 95 mmHg, confirmed on 2 separate visits before inclusion.
19. Heart rate in supine > 100 beats/min after 5 minute rest or untreated symptomatic bradycardia within one month prior to inclusion.
20. Total bilirubin > 1.5 times ULN, or ALT or AST > 3 times ULN.
21. Estimated GFR > 30 ml/min/1.73 m2 calculated by the modification of diet in renal disease (RD).
22. Chronic treatment with NSAIDs (> 7 days), except aspirin < 325 mg dose.
23. Uncontrolled insulin-dependent diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The efficiency of sodium excretion | 24 hours
  Will be assessed as the ratio between the average drug-induced natriuresis and the average drug recovered in urine over 24 hours.

SECONDARY OUTCOMES:
Pharmacokinetic plasma parameters and pharmacokinetic urine parameters | 24 hours
  Pharmacokinetic plasma parameters (Cmax, AUC0-t, AUC0-∞, t ½, Vd / F, Cl / F), pharmacokinetic urine parameters (ERFco , Ae24h, Ae ∞) and urine pharmacodynamic variables will be presented descriptively with no formal statistical testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigació de Medicaments (CIM), Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Ballester MR, Roig E, Gich I, Puntes M, Delgadillo J, Santos B, Antonijoan RM. Randomized, open-label, blinded-endpoint, crossover, single-dose study to compare the pharmacodynamics of torasemide-PR 10 mg, torasemide-IR 10 mg, and furosemide-IR 40 mg, in patients with chronic heart failure. Drug Des Devel Ther. 2015 Aug 5;9:4291-302. doi: 10.2147/DDDT.S86300. eCollection 2015. PMID 26273191